CLINICAL TRIAL: NCT02053844
Title: Analyzing the Impact of the Now iKnow Health Care Price Transparency Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alison Galbraith (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Bureau of Economic Research, Inc. (Other); Harvard Pilgrim Health Care (Other); Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor-Investigator, Alison Galbraith, Assistant Professor, Harvard Pilgrim Health Care
Organization: Harvard Pilgrim Health Care (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 5P30AG012810-20 (NIH); 5P01AG005842-27 (NIH)
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: no Specific Condition Targeted; Use of a Price Transparency Tool
Keywords: health care costs; quality of health care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- lottery and enhanced promotion of tool (Experimental): tool users in the intervention arm will be eligible to enter a monthly lottery to win one of two monthly drawings of a $500 gift card, and will receive enhanced promotion of the tool (mailed promotion, promotional message on the member web portal, and promotion through employers to employees)
  Interventions: Other: lottery for tool users to win a $500 prize; Other: enhanced promotion of the tool to employers and members
- usual promotion of the tool (No Intervention): Routine promotion of the tool through newsletter and on health plan web site

INTERVENTIONS:
Other: lottery for tool users to win a $500 prize — Intervention group is eligible to enter a monthly lottery to win a $500 gift card if they use the tool each month.
  Arms: lottery and enhanced promotion of tool
Other: enhanced promotion of the tool to employers and members — Intervention group also receives extra promotion of the tool through mailings, employer outreach, and automated phone calls
  Arms: lottery and enhanced promotion of tool

SUMMARY:
This project aims to assess the impact of a web-based health care cost and quality tool that is being implemented by a health plan for its members. The study will focus on members working for medium to large employers that have more than 90% of employees enrolled in deductible and tiered network health plans. The study will use an interrupted time series (ITS) design that includes random allocation of half of these employers to a study arm that will receive enhanced promotion of the tool and a $500 lottery incentive for its use in order to increase take-up. With these two study groups (a "high-dose" group receiving enhanced promotion and a lottery, and a "low-dose" group receiving routine promotion of the tool), the study will be able to evaluate whether access to a price transparency tool leads to reduced costs and more value-driven member behavior, and whether extra promotion increases take-up.

Members in the high-dose group who use the tool will be eligible to enter a monthly lottery to win a $500 prize during the 12-month intervention period. In addition to the lottery, employers in the high-dose group will receive additional promotional strategies such as a mailing and messages through the plan's member web portal to promote the tool and the lottery, and e-mails and flyers for employers to promote the tool and lottery to employees.

The aims of this project are to: 1) examine take-up of the tool and factors that predict take-up; and 2) to examine the impact of the tool on total and out-of-pocket health care costs and utilization

ELIGIBILITY:
Inclusion Criteria:

Health plan members from employers with at least 40 subscribers, of which at least 90% are currently in deductible plans or tiered network plans, and of which at least 80% were in deductible or tiered network plans in the prior year

Exclusion Criteria:

Members in non-group accounts and members in Medicare plans; members in states outside Massachusetts, New Hampshire, or Maine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81000 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
mean per-member-per-month total health care costs | monthly for 12 months
  employer level per-member-per-month total costs based on claims data

SECONDARY OUTCOMES:
percent of subjects using the tool | measured quarterly for 12 months
  Based on tool usage tracking data
mean per-member-per-month out-of-pocket costs | monthly for 12 months
  employer level per-member-per-month out-of-pocket costs based on claims data
per-member-per-month utilization of health care services | monthly for 12 months
  Employer-level utilization of health services based on claims data, including emergency department visits, encounters, lab services, radiology services, inpatient hospitalizations, MRIs, prescriptions

OTHER OUTCOMES:
reasons for using the tool | measured with each use of the tool, over 12 months
  based on survey report

CONTACTS AND LOCATIONS:
Overall Officials: Alison Galbraith, MD, MPH, Study Director — Harvard Pilgrim Health Care Institute and Harvard Medical Schooll; Jonathan Gruber, PhD, Principal Investigator — Massachusetts Institute of Technology
Locations (1):
- Harvard Pilgrim Health Care, Wellesley, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No